CLINICAL TRIAL: NCT06184139
Title: Effect of Maternal Age and BMI on Induction of Labor Using Oral Misoprostol in Late-term Pregnancies: a Retrospective Cross-sectional Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Andrea Etrusco, Principal investigator, University of Palermo
Other Study IDs: MISO-LATE_PREG
Record Dates: First submitted 2023-11-18; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Induction of Labor Affected Fetus / Newborn; Pregnancy Late
Keywords: Late-term pregnancy; body mass index; age; oral misoprostol; cervical ripening; induction of labor
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Misoprostol — Oral misoprostol for induction of labor in late term pregnancies

SUMMARY:
To evaluate the effect of maternal age and body mass index (BMI) on oral misoprostol induction of labor for late-term pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Late term pregnancies out of labor,
* Bishop score < 7

Exclusion Criteria:

* labor (defined as presence of at least three painful uterine contractions every ten minutes),
* uterine tachysystole (>5 contractions within 10 minutes for two consecutive 10-minute periods),
* hypertonic uterus,
* abnormal CTG,
* contraindications to vaginal delivery (fetal malpresentation such as breech presentation or transverse situation, fetal macrosomia, abnormally implanted placenta, active genital herpes infection, cervical cancer),
* patients with parity > 4,
* medical contraindication to misoprostol (asthma, glaucoma),
* women with previous hysterotomies.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: term (37 weeks or more of gestation) singleton pregnancies in women who have not had a previous cesarean delivery and a bishop score < 7.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of misoprostol for induction of labor | 290 days of pregnancy
  Efficacy induction of labor for late term pregnancies according to age and BMI

CONTACTS AND LOCATIONS:
Locations (1):
- Andrea Etrusco, Palermo, Italy